CLINICAL TRIAL: NCT00641784
Title: A Randomized Trial of Oral Nifedipine Versus Intravenous Magnesium Sulfate in the Acute Management of Preterm Labor in Women With Singleton Gestations, Intact Fetal Membranes, and Positive Vaginal Fetal Fibronectin
Brief Title: Tocolytics Trial: Intravenous (IV) Magnesium Versus Oral Nifedpine in Fetal Fibronectin (FFN) Postive Population
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: MemorialCare (Other)
Responsible Party: Kenneth Chan, Obstetrix (Magella)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 464-07
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Labor, Premature
Keywords: Composite Early neonatal Outcome; Late Neurological neonatal outcome
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral Nifedine
  Interventions: Drug: Nifedlipine
- 2 (Active Comparator): Intravenous Magnesium
  Interventions: Drug: Magnesium

INTERVENTIONS:
Drug: Magnesium — Intravenous Magnesium 6 gram load, 3 grams/hr
  Arms: 2
Drug: Nifedlipine — Oral Nifedpine 10 mgs q 20 min to effect (max 40mgs)...then 20 mgs q 4hrs
  Arms: 1

SUMMARY:
In women with singleton gestations, to contemporarily assess the efficacy of oral nifedipine versus intravenous magnesium sulfate in the acute management of preterm labor in terms of defined early and late neonatal measures

ELIGIBILITY:
Inclusion Criteria:

* Patients between 240/7-320/7 weeks gestation with findings consistent with preterm labor defined by at least one of the following criteria in accordance with regular uterine contractions (>4 uterine contractions in 20 minutes):

  1. Cervix > 2 cm in dilation or 80% effaced
  2. Positive fetal fibronectin (if performed).
  3. Demonstrated cervical change between two exams within 90 minutes.

Exclusion Criteria:

* Negative fetal fibronectin
* > 5cm dilatation
* Multiple gestations
* Known fetal anomalies or chromosomal abnormalities
* Ruptured membranes
* Significant vaginal bleeding
* Suspected chorioamnionitis
* Preeclampsia or uncontrolled hypertension
* Non-reassuring fetal heart tracing
* Placenta previa and/or accreta
* Placenta abruption
* Intrauterine growth restriction
* Maternal renal disease
* Underlying maternal cardiac condition
* Symptomatic hyperthyroidism
* Significant maternal disease
* Contraindication to nifedipine or magnesium
* Cerclage presence
* Tocolytic use within the last 12 hours
* Hypotension (defined as average blood pressure of <70/40's unresponsive to 1000 cc fluid bolus

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
In women with singleton gestations, to contemporarily assess the efficacy of oral nifedipine versus intravenous magnesium sulfate in the acute management of preterm labor in terms of defined early and late neonatal measures | At delivery

SECONDARY OUTCOMES:
To assess the efficacy of nifedipine versus intravenous magnesium in prolonging pregnancy in patients presenting with strict criteria of preterm labor. | At Delivery
To assess tolerance and side effects of nifedipine versus intravenous magnesium sulfate. | At delivery
To compare the total cost of using nifedipine versus intravenous magnesium sulfate in an acute hospital setting for tocolysis | At discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chan, MD, Principal Investigator — Obstetrix/Memorial Care; Vineet K Shrivastava, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Memorial Care Center for Women/Long Beach Memorial Medical Center, Long Beach, California, United States

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046